CLINICAL TRIAL: NCT00311051
Title: A Randomized Double-blind and Placebo-controlled Study to the Influence of Ramatroban/Montelukast Versus Montelukast/Placebo on the Early Allergic Reaction in Patients With Mild to Moderate Atopic Asthma (House Dust Mite)
Brief Title: Ramatroban/Montelukast Versus Montelukast/Placebo on the Early Allergic Reaction in Asthma Sensitive to House Dust Mite
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Research Center Borstel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAMONA-4022229; 4022229; Bundesinstitut (BfArM)
Record Dates: First submitted 2006-04-01; First posted 2006-04-05 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: Asthma; Allergens; house dust mites; Ramatroban; Montelukast; Bronchial Provocation Tests
MeSH Terms: conditions — Asthma | interventions — ramatroban; montelukast

INTERVENTIONS:
Drug: ramatroban
Drug: montelukast

SUMMARY:
The purpose of this study is to examine wether the combination of Ramatroban/Montelukast is as effective as Montelukast alone in patients with mild to moderate atopic asthma (GINA I and II) sensitive to house dust mite. The test is performed by a specific inhalative provocation.

DETAILED DESCRIPTION:
In the early allergic response in asthma, allergens connect to IgE on mast cells and basophile granulocytes. For that there are 3 main pathways in activation:

Besides quick liberation of Histamine and induction of cytokines there is a liberation of mediators from the arachidonate metabolism. In addition to Histamine there are especially Prostaglandin PGD2, Leukotriene LTC4 and also Thromboxane A2 for the classic symptoms of the early allergic reaction responsible. All of those mediators have potent bronchoconstrictive activity.

Prostaglandin D2 and Thromboxane A2 work on Thromboxane receptors. LTC4 links to Cys-LT-receptors.

According to an in-vitro-model of the early allergic reaction in human precision-cut lung slices with passive specific sensitization against grass-pollen, it has been shown that the early allergic response can only be suppressed partly by giving Antihistamines, Leukotriene receptor antagonists or Thromboxane receptor antagonist all on its own. It goes in consent with clinical findings, that all of these drugs alone have just an insufficient activity on asthma.

In the described human in-vitro-model the combination of Thromboxane receptor antagonist with Leukotriene receptor antagonist (Montelukast) blocked the early response in asthma completely.

These findings are the rationale for our study because so far there is no clinical data about the effect of the combination of Leukotriene receptor antagonist (Montelukast) with Thromboxane receptor antagonist.

The drug Montelukast is a Leukotriene receptor antagonist which is known for the treatment of mild to moderate asthma in Germany. According to the GINA-Guidelines Montelukast is given in addition to steroids and β-mimetics in asthma severity grade II and III.

The drug Ramatroban is a Thromboxane A2 receptor antagonist which is in Japan allowed for the treatment of allergic rhinitis. It also has an anti-asthmatic effect because it blocks bronchoconstriction, hyperresponsiveness of the airways and infiltration of inflammation cells. Furthermore, it has positive effects on allergic rhinitis by blocking the permeability of capillaries, blocking the nasal hyperresponsiveness and the infiltration of the mucosa by eosinophils.

During the studies Ramatroban has proved to be a save drug for the indication allergic rhinitis and also allergic asthma. In contrast to sufficient effectiveness in the indication allergic rhinitis it has been said that there is just insufficient effectiveness in the indication asthma.

About the combination of Ramatroban and Montelukast exists no clinical data so the study at hand examines the effect of Ramatroban/Montelukast versus Montelukast/Placebo on the early allergic reaction in patients with mild to moderate atopic asthma (GINA I and II) sensitive to house dust mites in a specific inhalative provocation.

ELIGIBILITY:
Inclusion Criteria:

* Atopic (house dust mite) asthma
* Severity GINA one and two

Exclusion Criteria:

* No reaction in specific bronchial provocation test
* Other kind of clinical relevant atopic reaction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Lung function by spirometry
Allergen concentration for specific bronchoprovocation

SECONDARY OUTCOMES:
Blood level of thromboxane and leukotriene metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zabel, Prof., Principal Investigator — Research Center Borstel
Locations (1):
- Research Center Borstel, Borstel, Germany

REFERENCES:
- [Background] Wohlsen A, Martin C, Vollmer E, Branscheid D, Magnussen H, Becker WM, Lepp U, Uhlig S. The early allergic response in small airways of human precision-cut lung slices. Eur Respir J. 2003 Jun;21(6):1024-32. doi: 10.1183/09031936.03.00027502. PMID 12797499